CLINICAL TRIAL: NCT01056562
Title: Testosterone-Guided Schedule of Androgen Deprivation Therapy (ADT) as an Alternative to A Fixed Schedule In Management Of Prostate Cancer
Brief Title: An Alternative to A Fixed Schedule In Management Of Prostate Cancer
Acronym: TADS
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: REB # 09-0526-C; NCT01007825 (obsolete NCT alias)
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Prostate Cancer
Keywords: Prostate; GU; Urological Oncology
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The male sex-hormone called testosterone is known to play a key role in the growth of prostate cancer. The usual treatment for the disease involves suppression of hormones (testosterone) by anti-hormonal treatment for an unknown period of time until the cancer progresses. This anti-hormonal treatment usually consists of injections every three months with an LHRH(Leutinizing Hormone-Releasing Hormone) agonist and a short course of anti-androgen pills, which together help to lower the production of testosterone. Long-term hormonal treatment has potentially serious side effects and is expensive.

In this study, hormonal treatments will be with held from those patients eligible and willing to participate. The aim of this study is to see if we can decrease the amount of hormone injections that patients require. This might lead to a decreased side effects(such as decrease in bone health, cardiovascular problems and metabolic syndrome which occurs when several health conditions happen at the same time and can lead to an increased risk of heart disease, stroke and diabetes) as well as to decrease the cost of hormonal therapy to treat prostate cancer.

DETAILED DESCRIPTION:
Most men respond to initial ADT with a fall in serum PSA and improvement in symptoms, if present initially; the median duration of response is about 1.5 - 2 years, but is highly variable. Increase in serum PSA despite a castrate testosterone level signifies that the disease has become castration resistant. Some patients may have short periods of response to other hormonal manipulations such as adding a peripheral antiandrogen such as bicalutamide, and later withdrawing it. Other hormonal manipulations may be tried sequentially before or after chemotherapy with varying success: this tertiary hormonal manipulation may include glucocorticoids such as prednisone or dexamethasone, ketoconazole and hydrocortisione, estrogens such as DES, and alternative anti-androgens such as flutamide and nilutamide. In most institutions, the policy is to continue the LHRH agonist indefinitely. Despite its proven role in prostate cancer treatment, ADT has multiple toxicities which include osteopenia/osteoporosis, a potentially lethal metabolic syndrome and cardiovascular complications. Also, continuous long term LHRH injections are very expensive.

In this study, we propose a prospective cohort study at Princess Margaret Hospital to answer the following important questions regarding tertiary hormonal manipulations:

1. What is the relationship between serum testosterone and time after stopping an LHRH agonist in men who have received chronic LHRH therapy for ≥ 1 year?
2. What clinical factors influence recovery of testosterone?
3. What is the saving of cost achieved by dosing the LHRH agonist on the basis of measurement of testosterone as compared to routine 3-monthly injection?

ELIGIBILITY:
Inclusion Criteria:

* Pathological evidence of adenocarcinoma of the prostate
* Have been Receiving an LHRH agonist (in the form of a 3-monthly depot) for at least 12 months
* Serum testosterone level below 1.5 nMol/L (≈43 mg/dl)

Exclusion Criteria:

* Patients on other clinical trials needing continuous androgen deprivation

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men with prostate cancer attending ambulatory clinics at Princess Margaret Hospital
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2009-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
We will monitor serum testosterone initially q 6 weeks increasing to every three months and delay initiating the next dose of ADT until serum testosterone level rises above 1.5nMol/l. | Baseline, Q6wks x 24 wks

SECONDARY OUTCOMES:
Jamar Dynamometer | Baseline and 18 weeks
EPIC Quality of Life Questionnaire | Baseline and 18 weeks
Six Minute Walk Test | Baseline and 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ian F Tannock, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada